CLINICAL TRIAL: NCT05733130
Title: Registro Italiano Pancreatite Cronica
Brief Title: Italian Registry Chronic Pancreatitis
Acronym: ITARECIPE
Status: Recruiting | Type: Observational
Sponsor: Associazione Italiana per lo Studio del Pancreas (Other)
Responsible Party: Sponsor
Other Study IDs: ITARECIPE
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Chronic Pancreatitis
Keywords: chronic pancreatitis; surveillance chronic pancreatitis; chronic pancreatitis diagnosis; chronic pancreatitis therapy
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ITARECIPE is a multicenter national registry designed to study the diagnosis and evolution of Chronic Pancreatitis

DETAILED DESCRIPTION:
Chronic pancreatitis (PC) is a relatively rare disease (45/100,000 population) in Italy, with heterogeneous aetiology, clinical history and treatment.

Patients need to be treated by different specialists, but almost always the gastroenterologist is central in diagnosis and treatment.

The study will be the first National Registry, prospective and will collect data on the history of the disease and its outcomes.

Data will be collected through an electronic data collection form (e-CRF) that the Sponsor (AISP) will make available to the Participating Centres.

Patients enrolled will be both new diagnoses or follow-up visits of patients with a diagnosis already made no more than 1 year before the signing of informed consent for the study in question: only data on the diagnosis and follow-up visits prior to the signing of the informed consent will be collected retrospectively (no more than one year).

Data from patients visited in the Centres included in the study will be collected prospectively.

In addition to the first visits, data will also be collected on follow-up visits that are scheduled according to the clinical need of each patient, which differ according to the stage of the disease

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 12 years;
* Diagnosis "definite" or "probable" according to the "M-ANNHEIM" criteria;
* First evidence of diagnosis within 12 months of enrolment.

Exclusion Criteria:

* Age < 12 years;
* History of known disease with certainty for > 12 months.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with:
  * a new suspected (both clinical and/or diagnostic evaluation, indicating a suspected diagnosis according to standard criteria)
  * established diagnosis of Chronic Pancreatitis and willing to provide their clinical and anamnestic information.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease Progression | 5 years
  The collection of data on disease progression in terms of the need for medical, endoscopic or surgical therapy, the risk of pancreatic exo-endocrine failure and the risk of developing pancreatic and extrapancreatic complications and death.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

REFERENCES:
- [Result] Olesen SS, Nojgaard C, Poulsen JL, Haas SL, Vujasinovic M, Lohr M, Lindkvist B, Bexander L, Gulbinas A, Kalaitzakis E, Ebrahim M, Erchinger F, Engjom T, Roug S, Novovic S, Hauge T, Waage A, Laukkarinen J, Parhiala M, Pukitis A, Ozola-Zalite I, Drewes AM; Scandinavian Baltic Pancreatic Club. Chronic Pancreatitis Is Characterized by Distinct Complication Clusters That Associate With Etiological Risk Factors. Am J Gastroenterol. 2019 Apr;114(4):656-664. doi: 10.14309/ajg.0000000000000147. PMID 30741740
- [Result] Engjom T, Nordaas IK, Tjora E, Dimcevski G, Haldorsen IS, Olesen SS, Drewes AM, Zviniene K, Barauskas G, Riis Jespersen HS, Jensen N, Borch A, Nojgaard C, Novovic S, Kardasheva SS, Okhlobystin A, Hauge T, Waage A, Frokjaer JB. Aetiological risk factors are associated with distinct imaging findings in patients with chronic pancreatitis: A study of 959 cases from the Scandinavian Baltic Pancreatic Club (SBPC) imaging database. Pancreatology. 2021 Jun;21(4):688-697. doi: 10.1016/j.pan.2021.02.023. Epub 2021 Mar 3. PMID 33707113
- [Result] Lohr JM, Dominguez-Munoz E, Rosendahl J, Besselink M, Mayerle J, Lerch MM, Haas S, Akisik F, Kartalis N, Iglesias-Garcia J, Keller J, Boermeester M, Werner J, Dumonceau JM, Fockens P, Drewes A, Ceyhan G, Lindkvist B, Drenth J, Ewald N, Hardt P, de Madaria E, Witt H, Schneider A, Manfredi R, Brondum FJ, Rudolf S, Bollen T, Bruno M; HaPanEU/UEG Working Group. United European Gastroenterology evidence-based guidelines for the diagnosis and therapy of chronic pancreatitis (HaPanEU). United European Gastroenterol J. 2017 Mar;5(2):153-199. doi: 10.1177/2050640616684695. Epub 2017 Jan 16. PMID 28344786
- [Result] Vege SS, Chari ST. Chronic Pancreatitis. N Engl J Med. 2022 Mar 3;386(9):869-878. doi: 10.1056/NEJMcp1809396. No abstract available. PMID 35235728
- [Result] de Rijk FE, Kempeneers MA, Bruno MJ, Besselink MG, van Goor H, Boermeester MA, van Geenen EJ, van Hooft JE, van Santvoort HC, Verdonk RC; Dutch Pancreatitis Study Group. Suboptimal care for chronic pancreatitis patients revealed by moderate to low adherence to the United European Gastroenterology evidence-based guidelines (HaPanEU): A Netherlands nationwide analysis. United European Gastroenterol J. 2020 Aug;8(7):764-774. doi: 10.1177/2050640620937610. Epub 2020 Jun 26. PMID 32588790
- [Result] Gardner TB, Adler DG, Forsmark CE, Sauer BG, Taylor JR, Whitcomb DC. ACG Clinical Guideline: Chronic Pancreatitis. Am J Gastroenterol. 2020 Mar;115(3):322-339. doi: 10.14309/ajg.0000000000000535. PMID 32022720
- [Result] Beyer G, Mahajan UM, Budde C, Bulla TJ, Kohlmann T, Kuhlmann L, Schutte K, Aghdassi AA, Weber E, Weiss FU, Drewes AM, Olesen SS, Lerch MM, Mayerle J. Development and Validation of a Chronic Pancreatitis Prognosis Score in 2 Independent Cohorts. Gastroenterology. 2017 Dec;153(6):1544-1554.e2. doi: 10.1053/j.gastro.2017.08.073. Epub 2017 Sep 14. PMID 28918191
- [Derived] Rizzo GEM, Apadula L, Piciucchi M, Stigliano S, Belfiori G, de Pretis N, Gabbrielli A, Barresi L, Frulloni L, Falconi M, Carrara S, Fabbri C, Capurso G; ITARECIPE study group. Italian Chronic Pancreatitis Registry (ITARECIPE): protocol for a nationwide cohort study. BMJ Open Gastroenterol. 2025 Apr 22;12(1):e001747. doi: 10.1136/bmjgast-2025-001747. PMID 40262909